CLINICAL TRIAL: NCT06434064
Title: A Pilot, Single-Arm, Phase II Trial of Tamoxifen Plus Pegylated Liposomal Doxorubicin in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Tamoxifen and Pegylated Liposomal Doxorubicin for the Treatment of Patients With Metastatic or Inoperable, Locally Advanced Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3671523; NCI-2024-03909 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3671523 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Unresectable Triple-Negative Breast Carcinoma; Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; liposomal doxorubicin; Doxorubicin; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (tamoxifen, pegylated liposomal doxorubicin) (Experimental): Patients receive tamoxifen PO QD on days 1-28 of each cycle and pegylated liposomal doxorubicin IV on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography, CT scan or MRI, tumor biopsy, and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Magnetic Resonance Imaging; Drug: Pegylated Liposomal Doxorubicin Hydrochloride; Drug: Tamoxifen

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; Dox-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; Doxorubicin Hydrochloride Liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; Liposomal Doxorubicin Hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; Pegylated Liposomal Doxorubicin; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99
Drug: Tamoxifen — Given PO
  Other Names: TMX

SUMMARY:
This phase II trial tests how well tamoxifen and pegylated liposomal doxorubicin works in treating patients with triple negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic) or that has spread to nearby tissue or lymph nodes (locally advanced) and is unable to be operated on (inoperable). Tamoxifen works by blocking the effects of estrogen in the breast. This may help stop the growth of tumor cells that need estrogen to grow. Doxorubicin is in a class of medications called anthracyclines. Doxorubicin damages the cell's DNA and may kill cancer cells. It also blocks a certain enzyme needed for cell division and DNA repair. Liposomal doxorubicin is a form of the anticancer drug doxorubicin that is contained inside very tiny, fat-like particles. Liposomal doxorubicin may have fewer side effects and work better than other forms of the drug. Giving tamoxifen and pegylated liposomal doxorubicin together may work better in treating patients with metastatic or inoperable, locally advanced triple negative breast cancer than giving either of these drugs alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of the combination of tamoxifen and pegylated liposomal doxorubicin in patients with metastatic or inoperable locally advanced triple negative breast cancer (TNBC) (estrogen receptor [ER] < 10%) as assessed by overall response rate (ORR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of pegylated liposomal doxorubicin given in combination with tamoxifen.

II. To determine clinical benefit including overall and progression free survival (overall survival [OS] and progression free survival [PFS]) as defined by RECIST v1.1.

III. To determine the duration of response.

EXPLORATORY OBJECTIVES:

I. To analyze changes in circulating tumor deoxyribonucleic acid (ctDNA) from longitudinal liquid biopsy to follow therapeutic response.

II. To determine estrogen receptor beta (ERβ)-mutant p53 interaction in tumors with in situ proximity ligation assay (PLA).

III. To analyze changes in gene expression by global ribonucleic acid (RNA)-sequencing (seq).

IV. To determine changes in the tumor microenvironment (TME) of tumors in response to treatment by analyzing tumor infiltrating lymphocytes (TILS) selected markers in the tumor and stromal tissues combined with CYBERSORT analysis of the transcriptome data.

V. Analyze changes in immune cell populations and circulating protein biomarkers as detectable from blood.

OUTLINE:

Patients receive tamoxifen orally (PO) once daily (QD) on days 1-28 of each cycle and pegylated liposomal doxorubicin intravenously (IV) on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography, computed tomography (CT) scan or magnetic resonance imaging (MRI), tumor biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed metastatic triple negative breast cancer (ER ≤ 10%) that have been previously treated with at least 2 lines of therapy in the metastatic setting
* Patients must have a confirmed eligible TP53 genomic alteration, as determined by the Roswell Park Oncomine™ Precision Assay (OPA) or similar CLIA-approved assay, using either an archival metastatic tumor sample or, if unavailable, a fresh biopsy. Uncertainty about the eligibility of the TP53 genomic alteration for this study can be resolved by discussion with the study PI
* Patients must have ERα (estrogen receptor alpha) and PgR (progesterone receptor) status assessed using current American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines. Patients are eligible if the tumor staining is ERα low/negative (ER ≤ 10%) and PgR negative by ASCO/CAP guidelines
* The tumor must be HER-2 negative by immunochemistry (IHC) 0-1+ or IHC 2 + and fluorescence in situ hybridization (FISH) negative
* Patients must be ≥ 18 years of age
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absolute neutrophil count (ANC) ≥ 1500/ μL
* Hemoglobulin (hb) ≥ 9 g/dL
* Platelet count ≥ 100,000/ μL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2 x ULN
* Creatinine clearance > 60 mL/min (Cockroft-Gault Equation)
* Left ventricular ejection fraction (LVEF) assessment must be performed within 30 days prior to enrollment. (LVEF assessment performed by 2-D echocardiogram is preferred; however, multigated acquisition scan [MUGA] scan may be substituted based on institutional preferences). The LVEF must be ≥ 50% regardless of the cardiac imaging facility's lower limit of normal
* Patients must be able to swallow oral medications
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients must not have any known contraindications to endocrine therapy, in the opinion of the treating investigator
* Participants who have had chemotherapy, hormonal/endocrine therapy, immunotherapy, biologics or radiotherapy (as well as any other investigational agents/devices) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to Cycle i Day 1 (6 weeks for nitrosoureas or mitomycin C), or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Have a known history of hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to tamoxifen or any of its excipients
* Patients known or suspected to have hypercoagulable syndrome or with history of venous or arterial thrombosis, stroke, transient ischemic attack (TIA), or pulmonary embolism
* Known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness
* Cardiac disease (history of and/or active disease) that would preclude the use of the drugs included in the treatment regimen. This includes angina pectoris, arrhythmias except for benign premature ventricular contractions, a history of myocardial infarction, documented congestive heart failure (CHF) or cardiomyopathy
* Patients with cirrhosis or severe hepatic impairment
* Patients must not have a condition or an uncontrolled intercurrent illness including, but not limited to any of the following: ongoing or active infection requiring systemic treatment, except uncomplicated urinary tract infection (UTI), or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 4 years
  Defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Will be summarized using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Incidence of adverse events | Until progression or end of treatment, up to 4 years
  Per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 will be summarized by attribution and grade using frequencies and relative frequencies.
Duration of response | From initial response to disease progression (per RECIST version1.1) up to 4 years
  Will be summarized using standard Kaplan-Meier methods, where the median times will be estimated with 90% confidence intervals.
Overall survival | From treatment initiation until death due to any cause, up to 4 years
  Will be summarized using standard Kaplan-Meier methods, where the median times will be estimated with 90% confidence intervals.
Progression free survival | From treatment initiation until disease progression or death due to any cause, up to 4 years
  Will be summarized using standard Kaplan-Meier methods, where the median times will be estimated with 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Sheheryar Kabraji, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States